CLINICAL TRIAL: NCT06401876
Title: Profiling Extracellular Vesicle Cargo in Obesity and Type 2 Diabetes
Brief Title: Extracellular Vesicle Cargo in Obesity and Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Temple University (Other)
Responsible Party: Principal Investigator, Michael A. Edwards, Principal Investigator, Mayo Clinic
Other Study IDs: 21-003883
Record Dates: First submitted 2024-05-02; First posted 2024-05-07 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Glucose Intolerance; Insulin Resistance; Diabetes
Keywords: Bariatric Surgical Procedure
MeSH Terms: conditions — Glucose Intolerance; Insulin Resistance; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of this research is to obtain blood samples before and after a bariatric procedure to better understand the reasons for glucose intolerance and insulin resistance (diabetes) in the obesity, and the reasons for improvement of diabetes after bariatric surgery

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in the Bariatric Surgery Program.
* Patients with A1c of 6.5 or higher within the last 6 months. OR
* Patients with A1c less than 6.5; have diagnosis of stable type 2 diabetes for > 6 months.

Exclusion Criteria:

* Disqualified for Bariatric Surgery.
* BMI < 35 kg/m^2.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is open to patients aged 21 years or older who have a BMI of 35 kg/m2 or more and are planning to undergo bariatric surgery. Patients must have an A1c of 6.5 or higher measured within the last 6 months or if A1C is less than 6.5 must have a diagnosis of stable type 2 diabetes for more than 6 months.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Identify circulating EV-derived protein and RNA signatures associated with T2D | 1 year
  Circulating EVs will be isolated from plasma samples from patients with extreme obesity, with either T2D or normoglycemia. EV-derived proteins will be analyzed by shotgun proteomics using mass spectrometry and RNA by sequencing or microarray RNA technology to identify differential abundance between T2D and normoglycemia.
Identify changes in circulating EV cargo in patients whose T2D resolves after sleeve gastrectomy (SG), Roux-en-Y gastric bypass (RYGB) or duodenal switch procedures. | 1 year
  Plasma samples will be prospectively obtained from patients recruited in Aim 1 at baseline and within four weeks and at one-year after SG, RYGB or Duodenal Switch Procedures. EVs will be isolated, and protein and RNA profiled as described in Aim 1. Changes in EV cargo from baseline to one-year post-SG or RYGB and T2D remission will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Edwards, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials